CLINICAL TRIAL: NCT03417947
Title: Vitamin D Intervention in Children With Sickle Cell Disease: A Pilot Randomized Controlled Trial
Brief Title: Vitamin D Supplementation in Children With Sickle Cell Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Euro-Pharm (Unknown)
Responsible Party: Principal Investigator, Genevieve Mailhot, Researcher, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ND
Record Dates: First submitted 2018-01-11; First posted 2018-01-31 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Sickle Cell Disease
Keywords: Bolus supplementation; Pilot randomised controlled trial; Vitamin D
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This is a randomised, quadruble-blind, placebo-controlled, parallel-group trial of vitamin D3 bolus supplementation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Applied Clinical Research Unit of Sainte-Justine UHC will generate the randomisation scheme. Group allocation codes will be held in a secure location with a restricted access by the Central pharmacy (Sainte-Justine UHC). All participants and research personnel, including the nurse, research trainee and research team will be blinded to group assignment.
  The supplier Euro-Pharm will provide the placebo and vitamin D3 preparations in coded bottles. Pharmacy will prepare the 6-mL bolus in coded syringes following the randomisation scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo identical to the vitamin D bolus in taste and appearance. The placebo will be administered once, at the beginning of the study. The oral liquid placebo will be prepared at the Pharmacy in coded syringes and will be administered to the participants by a nurse at the sickle cell disease Clinic.
  Interventions: Dietary Supplement: Placebo
- Vitamin D bolus (Experimental): The vitamin D bolus is an oral liquid supplement that will be administered once, at the beginning of the study. The oral liquid vitamin D bolus will be prepared at the Pharmacy in coded syringes and will be administered to the participants by a nurse at the sickle cell disease Clinic.The dose of vitamin D3 contained in the bolus is 300 000 IU.
  Interventions: Dietary Supplement: Vitamin D bolus

INTERVENTIONS:
Dietary Supplement: Vitamin D bolus — One single oral liquid vitamin D3 supplement of 300 000 IU
  Other Names: Cholecalciferol
  Arms: Vitamin D bolus
Dietary Supplement: Placebo — Placebo identical in taste and appearance to the vitamin D bolus
  Arms: Placebo

SUMMARY:
Sickle cell disease (SCD) is a genetic disease characterized by abnormal hemoglobin, the main constituent of red blood cells. People with SCD have nutritional deficiencies, and vitamin D deficiency is one of the most common. Symptoms of vitamin D deficiency are similar to those of SCD and include chronic pain and bone complications. Correcting vitamin D nutrition of children with SCD represents a treatment that will improve their health. A single oral high-dose of vitamin D3 will be given to SCD children during one of their follow-up visits at the SCD clinic of CHU Sainte-Justine, Montreal, Canada. This mode of administration was chosen to ensure a better adherence to the treatment. The investigators will determine whether this dose is safe and its administration feasible in clinic. The impact of this dose on blood vitamin D and calcium, urinary calcium, growth, inflammation, bone health, pain and quality of life will also be assessed. This study intends to propose a new intervention to improve the nutrition of children with this disease.

DETAILED DESCRIPTION:
Vitamin D deficiency is one of the most common nutritional conditions among patients with sickle cell disease (SCD). Since vitamin D deficiency and SCD share common manifestations including chronic pain, poor bone health and chronic systemic inflammation, it is reasonable to postulate that vitamin D deficiency may contribute to these complications. Thus, optimizing vitamin D nutrition represents an inexpensive strategy that may improve vitamin D status and health outcomes in SCD children. The working hypothesis is that administration of a single oral bolus of 300,000 IU of vitamin D3 to SCD children will result in the attainment of vitamin D sufficiency (25OHD levels >75 nmol/L) in 80% of participants after 3 months. The primary objectives are to assess feasibility, acceptability, and safety of the vitamin D3 bolus while secondary objectives are related to the mean change in serum 25OHD from baseline to 3 months post-bolus and its clinical impact. Seventy-two SCD children (5-17 years, SS and SC genotypes) will be randomized to one bolus of 300,000 IU of vitamin D3 or identical placebo. Blood will be collected at baseline and 3-month post-bolus to measure serum 25OHD and calculate the change from baseline at 3 months (efficacy outcomes). Other outcomes include urinary calcium/creatinine ratio and serum calcium (safety), questionnaires (acceptability and musculoskeletal pain) and parameters related to growth, haematology, inflammation and bone health (exploratory outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 5 and 17 years old who are followed up at the SCD Clinic, CHU Sainte-Justine, Montreal, Canada.

Exclusion Criteria:

* Conditions or use of medications known to interfere with calcium or vitamin D absorption or metabolism
* Known hypercalcemia
* Conditions characterized by a hypersensitivity to vitamin D (e.g. granulomatous disorders)
* Patients clinically diagnosed with rickets or other conditions requiring vitamin D therapy
* History or presence of urolithiasis
* Anticipated difficult follow up
* Patients already enrolled in other investigational studies
* Patients who have recently been hospitalized for severe pain crisis or acute sickle complication in the past 2 weeks
* Patients with unresolved pain issues

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Mean change in total serum 25-hydroxyvitamin D levels | 3 months
  Group difference in the mean change in total serum 25OHD from baseline to 3 months.

SECONDARY OUTCOMES:
Vitamin D sufficiency | 3 months
  Difference in the proportion of children with serum 25-hydroxyvitamin D ≥75nmol/L at 3 months

OTHER OUTCOMES:
Hypercalciuria | 7 days post-intervention
  Number of patients with urinary calcium to creatinine ratio above normal reference range for age
Hypercalcemia | 3 months
  Number of patients with serum calcium above normal reference range for age
Serum 25-hydroxyvitamin D levels | 3 months
  Number of patients with serum 25-hydroxyvitamin D levels >250 nmol/L
Mean change in weight | 3 months
  Group difference in the mean change of weight (kg) from baseline to 3 months.
Mean change in height | 3 months
  Group difference in the mean change of height (kg) from baseline to 3 months.
Mean change in hemoglobin | 3 months
  Group difference in the mean change of circulating hemoglobin from baseline to 3 months.
Mean change in fetal hemoglobin | 3 months
  Group difference in the mean change of circulating fetal hemoglobin from baseline to 3 months.
Mean change in leucocyte counts | 3 months
  Group difference in the mean change of blood leucocyte counts from baseline to 3 months.
Mean change in platelet counts | 3 months
  Group difference in the mean change of blood platelet counts from baseline to 3 months.
Mean change in reticulocyte counts | 3 months
  Group difference in the mean change of blood reticulocyte counts from baseline to 3 months
Mean change in neutrophil counts | 3 months
  Group difference in the mean change of blood neutrophil counts from baseline to 3 months
Mean change in mean corpuscular volume | 3 months
  Group difference in the mean change of blood mean corpuscular volume from baseline to 3 months
Mean change in serum creatinine | 3 months
  Group difference in the mean change of serum creatinine from baseline to 3 months.
Mean change in serum bilirubin | 3 months
  Group difference in mean change of serum bilirubin from baseline to 3 months.
Mean change in serum parathyroid hormone | 3 months
  Group difference in mean change of serum parathyroid hormone from baseline to 3 months
Mean change in serum P1NP | 3 months
  Group difference in mean change of serum amino-terminal propeptide of type I collagen (P1NP) from baseline to 3 months
Mean change in serum C-telopeptides | 3 months
  Group difference in mean change of serum C-telopeptides from baseline to 3 months
Mean change in musculoskeletal pain scores | 3 months
  Musculoskeletal pain will be assessed with the Brief Pain Inventory (BPI). Group difference in the mean change in BPI scores.
Mean change in quality of life scores | 3 months
  Health-related quality of life will be assessed through the Pediatric Quality of life (PedQoL) inventory. Group difference in the mean change in PedQoL scores.
Sickle cell disease-related complications | 3 months
  Occurrence of sickle cell disease complications affecting bone, the kidneys, the retina, blood vessels, the heart, the lungs, the spleen, the liver and gallbladder during the study period
Participant recruitment | 3 months
  Percentage of patients recruited from those screened
Participant retention | 3 months
  Percentage of patients retained for the entire study duration
Participant compliance | 3 months
  Percentage of patients who comply with the study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Mailhot, PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soe HHK, Abas AB, Than NN, Ni H, Singh J, Said ARBM, Osunkwo I. Vitamin D supplementation for sickle cell disease. Cochrane Database Syst Rev. 2020 May 28;5(5):CD010858. doi: 10.1002/14651858.CD010858.pub3. PMID 32462740

DOCUMENTS (1):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03417947/Prot_000.pdf